CLINICAL TRIAL: NCT03290443
Title: A Phase 1, Open-Label Single-Dose Study to Assess the Pharmacokinetics of Enasidenib (AG 221, CC 90007) in Subjects With Moderate and Severe Hepatic Impairment.
Brief Title: A Study to Assess the Pharmacokinetics of Enasidenib (CC-90007) in Subjects With Moderate and Severe Hepatic Impairment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90007-CP-003; U1111-1202-3186 (Registry Identifier: WHO)
Expanded Access: NCT03723057 (No longer available)
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Hepatic Impairment
Keywords: Hepatic; Pharmacokinetics; Phase 1; Enasidenib; CC-90007
MeSH Terms: interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enasidenib (CC-90007) tablet (Experimental): Subjects will receive one 100 mg enasidenib (CC-90007) tablet the morning of Day 1 which will be administered in the fasted state.
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — 100 mg enasidenib (CC-90007)
  Other Names: AG-221; AG-221 mesylate; AGI-12910; AGI-12910 mesylate; CC-90007, IDHIFA

SUMMARY:
This is a multi-center, open-label study to assess the PK of single 100 mg oral dose of enasidenib (CC-90007) in subjects with moderate and severe hepatic impairment, and in matched healthy control subjects with normal hepatic function.

Degrees of hepatic impairment will be determined during screening by the subject's score according to Pugh's Modification of Child's Classification of Severity of Liver Disease

DETAILED DESCRIPTION:
Subjects will be enrolled in Groups 1 through 4 as follows:

* Group 1: Approximately 6 to 8 male and female subjects with moderate hepatic impairment (with a Child-Pugh score of ≥ 7 to ≤ 9) will be enrolled in Group 1.
* Group 2: Approximately 6 to 8 healthy male and female subjects with normal hepatic function will be enrolled in Group 2. Subjects in Group 2 will be matched to subjects in Group 1 with respect to sex, age (± 10 years), and weight (± 30 pounds).
* Group 3: Approximately 6 to 8 male and female subjects with severe hepatic impairment (with a Child-Pugh score of ≥ 10 to ≤ 13) will be enrolled in Group 3.
* Group 4: Approximately 6 to 8 healthy male and female subjects with normal hepatic function will be enrolled in Group 4. Subjects in Group 4 will be matched to subjects in Group 3 with respect to sex, age (± 10 years), and weight (± 30 pounds). This study employs a staged design as follows.
* At least 4 subjects with moderate hepatic impairment must demonstrate satisfactory safety and tolerability for up to 8 days after dosing, before subjects with severe hepatic impairment may be dosed.
* Two subjects with severe hepatic impairment must demonstrate satisfactory safety and tolerability for up to 8 days after dosing, before the remaining subjects with severe hepatic impairment may be dosed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for all subjects (Group 1, 2, 3, and 4)

Each subject must satisfy all of the following criteria to be enrolled in the study:

Key inclusion criteria:

1. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject is male, or non-pregnant and non-nursing female between ≥ 40 and ≤ 65 years of age at the time of signing the ICF.
3. Subject has body mass index (BMI) ≥ 18 and ≤ 40 kg/m2 at screening.
4. Subject has seated systolic blood pressure (BP): 90 to 160 mmHg, seated diastolic BP: 50 to 100 mmHg, and pulse rate: 40 to 100 bpm.
5. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at screening).
6. Females of childbearing potential (FCBP)1 must have a negative pregnancy test at the Screening and Baseline Visits. While receiving IP and for at least 4 months after taking the last dose of IP, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options.
7. Male subjects must:

   a. Practice true abstinence2 (which must be reviewed on a monthly basis and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP while participating in the study, during dose interruptions, and for at least 4 months after the last dose of IP, even if he has undergone a successful vasectomy.

   Inclusion Criteria for Subjects with Moderate or Severe Hepatic Impairment (Groups 1 and 3) Each subject with moderate or severe renal impairment must also meet ALL of the criteria listed below for entry:
8. Subject has moderate or severe hepatic impairment or cirrhosis due to chronic hepatic disease and/or prior alcohol use.
9. Subject has moderate (Group 1), or severe (Group 3) hepatic impairment as defined by Child-Pugh Score.

   * Group 1 subjects must have moderate hepatic impairment and are required to have documentary confirmation of the diagnosis of cirrhosis made by biopsy, laparoscopy, or imaging study with a Child-Pugh score of ≥ 7 to ≤ 9, at screening.
   * Group 3 subjects must have severe hepatic impairment. If biopsy or laparoscopy is not performed prior to screening, subject can be included only if they have chronic liver disease and objective evidence of portal hypertension (ascites diagnosis by imaging or varices), or current medication for consequences of portal hypertension. In either case a Child-Pugh score of ≥ 10 to ≤ 13 at screening is required.
10. Subject has a normal or clinically acceptable 12-lead ECG at screening. In addition:

    • Subject (male or female) has a QTcF value ≤ 480 msec at screening.
11. Must be stable in concomitant medication regimen (defined as not starting a new medication[s] or a change in the dosage or frequency of the concomitant medication[s] within 7 days or 5 half-lives [whichever is longer] before dosing with study drug).
12. Subjects may be treated with diuretics for ascites; however, subjects with severe ascites at time of enrollment may only be included at the discretion of the investigator with agreement of the Sponsor.
13. Subjects may have a history of encephalopathy; however, they must be on stable treatment for at least 1 month prior to screening, and must not have had an acute encephalopathic episode in the 1 months prior to screening.
14. Subjects must not have history of hepatorenal syndrome or hemolysis. Inclusion Criteria for a Matched Healthy Subject (Groups 2 and 4)

    Each matched healthy subject must meet ALL the criteria listed below for entry:
15. Subject must be free of any clinically significant disease that would interfere with the study evaluations.
16. Subject must have liver-related laboratory test results within the respective reference ranges or with clinically insignificant excursions therefrom as agreed by the Investigator and Celgene's Medical Monitor.
17. Subject must match a subject in Group 1 or 3, as needed with respect to sex, age (± 10 years), and weight (± 30 pounds).
18. Subject must be in good health as determined by past medical history, PE, vital signs, ECG, and clinical laboratory safety tests. Clinical laboratory safety tests (ie, hematology, chemistry, and urinalysis) and 12-lead ECGs must be within normal limits or clinically acceptable as judged by the Investigator.
19. Subject has a normal or clinically acceptable 12-lead ECG at screening. In addition:

    1. If male, subject has a QTcF value ≤ 450 msec at screening.
    2. If female, subject has a QTcF value ≤ 470 msec at screening.

Exclusion Criteria:

Exclusion Criteria for all subjects (Groups 1, 2, 3, and 4)

The presence of any of the following will exclude a subject from enrollment:

Key exclusion criteria

1. Subject has any condition or circumstance that prevents the subject from understanding and signing the ICF.
2. Subject has any condition that places the subject at an unacceptable risk from participating in the study or would confound the ability to interpret data from the study.
3. Subject has any significant medical condition or psychiatric illness that would prevent the subject from participating in the study at Investigator discretion.
4. Subject has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, excretion, eg, bariatric procedure. Subjects with cholecystectomy and appendectomy may be included.
5. Subject is a pregnant or is breastfeeding.
6. Subject donated blood or plasma within 2 weeks before dose administration to a blood bank or blood donation center.
7. Subject has a history of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 6 months before the first dose administration, or positive alcohol screen.
8. Subject has a history of drug abuse (as defined by the current version of the DSM) within 6 months before the first dose administration, or positive drug screen that is not consistent with the patient's prescribed medication and or/medical history.
9. Subject is known to have active serum hepatitis, or have a positive result to the test for Human immunodeficiency virus (HIV) antibodies at screening.

   • Chronic or resolved Hepatitis B or Hepatitis C are acceptable only if sequelae are limited to hepatic involvement and its consequent comorbidities. (ie, vasculitis, clinically significant cryoglobulinemia, etc. are unacceptable).
10. Subject was exposed to an investigational drug (new chemical entity) within 30 days before dosing, or 5 half-lives of that investigational drug, if known (whichever is longer).
11. Subject used approved medications or herbal medicines that are moderate or strong cytochrome P450 (CYP)1A2 or 3A4/5 inducers and/or inhibitors (including St. John's wort) within 14 days or 5 half-lives of screening, whichever is longer.

    • The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inhibitors and/or inducers of CYP1A2 and CYP3A4/5.

    (http://medicine.iupui.edu/clinpharm/ddis/table.aspx).
12. Subject will have consumed Seville oranges, grapefruit or grapefruit juice and/or pomelos, exotic citrus fruits, or grapefruit hybrids within 14 days or 5 half-lives of dosing, whichever is longer.
13. Subject smokes more than 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
14. Subject has a history of multiple drug allergies or drug-related anaphylaxis.
15. Subject has received live vaccination (excluding seasonal flu vaccination) within 90 days of dosing.
16. Subject is part of the staff personnel or a family member of the investigational study staff.
17. Subject is, for any reason, deemed by the investigator to be inappropriate for this study, including a subjects who is unable to communicate or to cooperate with the investigator or the clinical staff. Exclusion Criteria for Subjects with Moderate or Severe Hepatic Impairment (Groups 1 and 3)

    The presence of any of the following will exclude a hepatic impaired subject from enrollment:
18. Subject has any unstable medical condition occurring within 3 months prior to signing the ICF (excluding hepatic impairment and associated comorbidities per Investigator discretion).
19. Subject has any serious medical condition (excluding hepatic impairment and related complications), clinically significant laboratory abnormality not related to hepatic impairment and related complications, or psychiatric illness that would prevent the subject from signing the ICF and participating in the study per Investigator discretion.
20. Subject has hepatic encephalopathy with time- or place- disorientation, somnolence, stupor, rigidity, coma, no personality/behavior, rigidity, or hyperactive reflexes - or has had such within 1 month of screening.
21. Subject has a history of incipient/planned liver transplantation within 6 months of screening or has received a liver transplant.

    Exclusion Criteria for a Matched Healthy Subject (Groups 2 and4)

    Each matched healthy subject will be excluded from entry if ANY of the criteria listed below are met:
22. Subject has any clinically significant laboratory abnormality that in the opinion of the Investigator, is considered to prevent the subject from safely completing the study.
23. Subject has any unstable clinically significant illness within 3 months prior to the study.
24. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
25. Positive testing for any active hepatitis, or history of Hepatitis B or C.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | Day 1
  Estimation of maximum observed plasma concentration
Pharmacokinetics - AUC0-∞ | Up to Day 36
  Estimation of AUC from time zero extrapolated to infinity
Pharmacokinetics - AUC0-t | Up to Day 36
  Estimation of AUC from time zero extrapolated to last time point
Pharmacokinetics - tmax | Day 1
  Time to reach Cmax

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene
Locations (5):
- United States (5):
  - DaVita Clinical Research, Lakewood, Colorado
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center OCRC, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - New Orleans Center of Clinical Research, Knoxville, Tennessee